CLINICAL TRIAL: NCT03714269
Title: Acute Effects of a Passive Stretching Session on the Mechanical Properties of Medial Gastrocnemius Muscle in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18CH121; ANSM (Other: 2018-A01921-54)
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2018-10

CONDITIONS: Cerebral Palsy
Keywords: children; medial gastrocnemius muscle
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Children with cerebral palsy of the spastic type (Experimental)
  Interventions: Other: measurement evaluated with an isokinetic dynamometer; Other: measurement evaluated with an 2D ultrasound; Other: assessment of the level of discomfort

INTERVENTIONS:
Other: measurement evaluated with an isokinetic dynamometer — measurement of the maximum dorsiflexion angle in degrees evaluated on an isokinetic dynamometer
Other: measurement evaluated with an 2D ultrasound — * simultaneous recording of force torque, joint angle and myotendinous junction displacement in 2D ultrasound during 5 passive mobilization cycles of ankle flexion-extension at very low speed
  * recording of static images in 2D ultrasound representing the proximal insertion of the gastrocnemius muscle in the internal condyle of the femur, the myotendinous junction.
Other: assessment of the level of discomfort — visual analogue scale (0 = no discomfort and 10 = maximal discomfort)

SUMMARY:
Children with cerebral palsy present early in the childhood altered muscular properties, as soon as structural or stiffness. In the gastrocnemius muscle, altered muscular properties are characterized by short muscle belly length and increased stiffness which contribute to contracture and limiting joint range of motion. This study assess efficacy of an acute high intensity and long-time stretching session of plantarflexors muscle on their viscoelasticity properties and maximal dorsiflexion angle gain. Single stretching session is characterized by high intensity and long time (5 minutes).

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy of the spastic type
* Children with a maximum dorsal ankle flexion amplitude limitation of less than 10°.

Exclusion Criteria:

* Children who have undergone surgery on the lower limbs.
* Children with a botulinum toxin injection and/or a series of elongation casts for less than three months.
* Children with ongoing analgesic treatment

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2018-11-28 (Actual); Study Completion 2018-11-28 (Actual)

PRIMARY OUTCOMES:
slope of the torque curve force-ankle joint angle in the joint area -25° plantar flexion/maximum dorsal flexion | baseline

SECONDARY OUTCOMES:
Maximum dorsal flexion angle of ankle, knee in maximum extension position | at 5 minutes
slope of the force-displacement torque curve myotendinous junction of the Sural Triceps in the articular sector -25° plantar flexion/maximum dorsal flexion | at 5 minutes
lengths of the musculotendinous unit of the Triceps Sural muscle, the muscular body of the gastrocnemius muscle and the Achilles tendon in cm measured at rest, knee in maximum extension position, ankle angle in neutral plantar/dorsal flexion position. | at 5 minutes
visual analogue scale of discomfort | at 5 minutes
  0 = not discomfort and 10 = maximal discomfort

CONTACTS AND LOCATIONS:
Overall Officials: Vincent GAUTHERON, Principal Investigator — CHU de Saint Etienne
Locations (1):
- CHU de Saint Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boulard C, Gautheron V, Lapole T. Acute passive stretching has no effect on gastrocnemius medialis stiffness in children with unilateral cerebral palsy. Eur J Appl Physiol. 2023 Mar;123(3):467-477. doi: 10.1007/s00421-022-05046-7. Epub 2022 Nov 1. PMID 36318307